CLINICAL TRIAL: NCT00975299
Title: Open-label, Multicenter PET/CT (Positron Emission Tomography/Computed Tomography) Study for Investigation of Safety, Tolerability, Biodistribution and Diagnostic Performance of the 18F Labeled PET Tracer BAY86-4367 Following a Single Intravenous Administration of 300 MBq (Corresponding to </= 40 µg Mass Dose) in Patients With Prostate Cancer as Well as Radiation Dosimetry, Plasma Pharmacokinetics, Biodistribution, Safety and Tolerability of the Tracer in PET/CT in Healthy Volunteers
Brief Title: Positron Emission Tomography/Computed Tomography (PET/CT) Imaging for Radiation Dosimetry, Plasma Pharmacokinetics, Biodistribution, Safety and Tolerability and Diagnostic Performance of BAY86-4367 in Patients With Prostate Cancer and Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13991; 2008-007460-42 (EudraCT Number)
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Diagnostic Imaging
Keywords: Neoplasm; PET/CT diagnosis; PET tracer
MeSH Terms: conditions — Neoplasms | interventions — BAY 86-4367

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-4367
- Arm 2 (Experimental)
  Interventions: Drug: BAY86-4367

INTERVENTIONS:
Drug: BAY86-4367 — Cancer patients, single intravenous bolus injection of 300 MBq BAY86-4367 on day one of the treatment period, PET/CT
  Arms: Arm 1
Drug: BAY86-4367 — Healthy volunteers, single intravenous bolus injection of 300 MBq BAY86-4367 on day one of the treatment period, whole body PET/CT for determination of effective dose., kinetics of BAY86-4367 in blood
  Arms: Arm 2

SUMMARY:
Visual assessment of diagnostic PET/CT (positron emission tomography/computed tomography) images obtained after a single intravenous injection of BAY86-4367 in patients with cancer

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

  * males, >/=50 and <= 65 years of age
* Cancer patients:

  * males >/= 45 years of age
  * patients with recurrent prostate cancer had a positive choline PET/CT for detection, or staging, or restaging of cancer, evaluation of the primary prostate cancer detection rate with BAY 86-4367 in comparison to histology as standard of truth (choline PET/CT is optional).

Exclusion Criteria:

* Exclusion criteria for all healthy volunteers and patients:

  * Concurrent severe and/or uncontrolled and/or unstable other medical disease (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 12 months prior to planned injection of BAY 86-4367, unstable and uncontrolled hypertension, chronic renal or hepatic disease, severe pulmonary disease) which could compromise participation in the study
  * Known sensitivity to the study drug or components of the preparation.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Visual assessment of lesions | Day of study drug administration

SECONDARY OUTCOMES:
Quantitative analysis of BAY86-4367 uptake into lesions (Standardized Uptake Values = SUVs) | Day of study drug administration
Electrocardiogram (ECG) | At least 3 times within 8 days after treatment
Blood pressure | At least 3 times within 8 days after treatment
Serum protein | At least 3 times within 8 days after treatment
Serum creatinine | At least 3 times within 8 days after treatment
Serum GOT (Glutamat-Oxalacetat-Transaminase) | At least 3 times within 8 days after treatment
Adverse events collection | At least 3 times within 8 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- München, Bavaria, Germany
- Zurich, Canton of Zurich, Switzerland